CLINICAL TRIAL: NCT01290770
Title: Search a Correlation Between Lipoprotein(a) Rate and TFPI(Tissue Factor Pathway Inhibitor)Activity in Obese Patients With Chest Pain Like Angina
Brief Title: Search a Correlation Between Lp(a) Rate and TFPI Activity in Obese Patients With Chest Pain Like Angina
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008178
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Atherosclerosis
Keywords: obesity; men; TFPI; Lipoprotein(a); Lp(a); Tissue Factor pathway inhibitor; aspirin
MeSH Terms: conditions — Atherosclerosis; Obesity; Multiple Endocrine Neoplasia Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese men: obese men with chest pain like angina
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sample at inclusion and 1 month after inclusion

SUMMARY:
Atherosclerotic cardiovascular disease is a leading cause of mortality in our countries. Clinically, symptoms could be chest pain suggesting stable angina. Atherosclerosis is influenced by cardiovascular risk factors which obesity (Body Mass Index>30). Obesity is associated with an increase risk of cardiovascular complications.

Lipoprotein(a) is regarded as an independent risk factor for premature cardiovascular disease. Lp(a) is composed of low-density lipoprotein - like particle bound to glycoprotein molecule: apolipoprotein(a). Plasma levels are determinated to more than 90% by genetic factors (no significant influence of statin, weight, lifestyle factor: diet, exercise). Two study with few patients have found that aspirin lowers serum Lp(a) levels. Elevated Lp(a) is a risk factor for recurrent coronary events in obese patient.

Atherosclerosis is associated with imbalance of coagulation. TFPI (tissue factor pathway inhibitor) is the earliest inhibitor of the blood coagulation process, natural direct inhibitor of tissue factor. In-vitro, TFPI activity is inhibited by high Lp(a) .

The aim of this study is to research reverse association between Lp(a) and TFPI activity in obese patient with chest pain like stable angina suggesting atherosclerotic heart disease and effect of aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Men
* Obese BMI>30
* No aspirin treatment before inclusion
* Coronary exploration: coronary angiography or tomography coronary angiography
* Chest pain like stable angina

Exclusion Criteria:

* Women
* Severe hepatic insufficiency
* Inflammatory disease
* Neoplasia
* Protein S deficiency
* Aspirin treatment 10 days before inclusion
* Oral anticoagulant treatment at inclusion
* Heparin or low molecular weight heparin treatment at inclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese men with chest pain like stable angina
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
correlation between Lp(a) and TFPI activity | day 1
  Establish correlation between Lp(a) rate and TFPI activity in obese patients with chest pain like stable angina

SECONDARY OUTCOMES:
Correlation between Lp(a) and TFPI resistance | day 1
  Establish correlation between Lp(a) rate and TFPI resistance at inclusion and 1 month after aspirin treatment
Correlation between lp(a) rate and TFPI activity | 1 month
  Establish the correlation, 1 month after initiation of aspirin treatment, between lp(a) rate and TFPI activity
thrombin generation | day 1
  describe thrombin generation with calibrated automated thrombinography technique in obese patient with chest pain like angina and hight Lp(a)rate
Correlation between Lp(a) and TFPI resistance | 1 month
  Establish correlation between Lp(a) rate and TFPI resistance at inclusion and 1 month after aspirin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte TARDY, MD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - Service de cardiologie - CHG Feurs, Feurs
  - Service de cardiologie - CHG Firminy, Firminy
  - Service de cardiologie - CHU de Saint-Etienne, Saint-Etienne